CLINICAL TRIAL: NCT01847469
Title: Zonisamide in Addition to Enhanced Cognitive Processing Therapy-C (E-CPT-C) for Veterans With PTSD and Comorbid Alcohol Dependence
Brief Title: Zonisamide in Addition to E-CPT-C for Veterans With PTSD and Comorbid Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ismene Petrakis, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1211011063; 01641 (Other: VA IRB)
Record Dates: First submitted 2013-01-23; First posted 2013-05-06 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Dependence; Post-Traumatic Stress Disorder (PTSD)
Keywords: Alcohol Dependence; Post-Traumatic Stress Disorder (PTSD); Zonisamide; Cognitive Processing Therapy (CPT)
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zonisamide (Experimental): Participants in this arm will receive zonisamide for 12 weeks.
  Interventions: Behavioral: Enhanced-Cognitive Processing Therapy-C (E-CPT-C); Drug: Zonisamide
- Placebo (Placebo Comparator): Participants in this arm will receive placebo medication for 12 weeks.
  Interventions: Behavioral: Enhanced-Cognitive Processing Therapy-C (E-CPT-C); Drug: Placebo

INTERVENTIONS:
Behavioral: Enhanced-Cognitive Processing Therapy-C (E-CPT-C)
Drug: Zonisamide
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, controlled trial with 50 veterans diagnosed with post-traumatic stress disorder (PTSD) and comorbid alcohol dependence. Veterans will be randomized to receive either zonisamide (400 mg) or placebo for 12 weeks in a double blind fashion. Randomization will be done using 3:1 ratio and will be performed by our research pharmacy using a random assignment in blocks of 4- 3 will be assigned to active medication and 1 to placebo. Medication will be titrated over a 6 week titration phase followed by a 6 week treatment phase. All veterans will receive E-CPT-C therapy for the 12 weeks of treatment; E-CPT-C will be provided by trained and qualified clinicians with extensive experience providing E-CPT-C. Veterans will be recruited primarily through advertisement, but also through the clinical facilities at the VA and from other collaborators.

ELIGIBILITY:
Inclusion Criteria:

* Current alcohol dependence, as determined by a structured clinical interview (Structured Clinical Interview for DSM-IV Axis I Disorders) (SCID)
* Current PTSD as determined by a structured clinical interview (SCID)
* Veterans with current alcohol dependence, with at least one recent episode of heavy drinking over the past 14 days.
* Medically and neurologically healthy on the basis of history, physical examination, EKG, screening laboratories
* For women, negative pregnancy test and use of acceptable method of contraception

Exclusion Criteria:

* Females who are pregnant or lactating.
* Veterans with a current unstable medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology, which in the opinion of the physician would preclude the subject from fully cooperating or be of potential harm during the course of the study
* Veterans who meet current SCID criteria for a major Axis I diagnosis (Bipolar Disorders, Schizophrenia and Schizophrenia-type Disorders).
* History of substance dependence (other than alcohol, tobacco or cannabis) by DSM-IV criteria in the last 90 days.
* Veterans taking mood stabilizers and antipsychotic medications for specific psychiatric disorders.
* Veterans with a history of allergy to zonisamide.
* Veterans already receiving CPT.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide: Participants in this arm will receive zonisamide for 12 weeks.
  Enhanced-Cognitive Processing Therapy-C (E-CPT-C)
  Zonisamide
- Placebo: Participants in this arm will receive placebo medication for 12 weeks.
  Enhanced-Cognitive Processing Therapy-C (E-CPT-C)
  Placebo
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 18 | 6
Completed | 9 | 3
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.28 (12.94) | 47.83 (11.57) | 45.17 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 4 | 22
  Male | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 3 | 10
  African American | 7 | 1 | 8
  Hispanic | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days
Description: Using a 90 day Timeline Follow Back (TLFB), the total number of drinking days at baseline and at 12 weeks of treatment were used.
Time Frame: 12 weeks
Population: The intention to treat population was used in the analysis.
Measure: Mean (Standard Error); unit: days
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 18 | 6
days
  Baseline | 46.87 (5.63) | 51.00 (9.48)
  12 weeks | 7.44 (5.47) | 17.33 (9.48)

2. Primary Outcome: Number of Heavy Drinking Days
Description: Timeline Follow Back (TLFB) will be used to document the number of "heavy" drinking days during 12 weeks of treatment. Heavy drinking is defined as greater than or equal to 5 drinks for men and greater than or equal to 4 drinks for women.
Time Frame: 12 weeks
Population: The intention to treat population was used in the analysis.
Measure: Mean (Standard Error); unit: days
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 18 | 6
days
  Baseline | 43.94 (5.37) | 31.50 (9.05)
  12 weeks | 5.50 (5.22) | 4.16 (9.05)

3. Primary Outcome: Clinician-Administered PTSD Scale (CAPS) Total Score
Description: The Clinician-Administered PTSD Scale (CAPS) Total Score will be used to measure PTSD symptoms at the end of the 12 week intervention. The CAPS Total Score is a summing of the 17 items that are each scored 0-4- where 0 indicates "none". The range of Total Scores can be 0 to 136, where 136 would be the highest amount of scored PTSD symptoms.
Time Frame: 12 weeks
Population: The intention to treat population was used in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 18 | 6
units on a scale
  Baseline | 67.33 (5.49) | 72.83 (9.51)
  12 weeks | 30.83 (6.02) | 23.80 (11.21)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were collected with a weekly questionnaire of side effects over the 12 week period.
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/6
Other Adverse Events (participants affected / at risk) | 6/18 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=18) | Placebo (N=6)
Suicidal Ideation (Psychiatric disorders) | 0 | 1 — Patient hospitalized due to intoxication and suicidal ideation.
Fall (General disorders) | 0 | 1 — Patient taken to emergency care following a fall.
Breast Swelling (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=18) | Placebo (N=6)
Difficulty Sleeping (General disorders) | 6 | 2
Depressed Mood (Psychiatric disorders) | 6 | 1
Fatigue (General disorders) | 3 | 1
Drowsiness (General disorders) | 3 | 1
Decreased Libido (Psychiatric disorders) | 3 | 2
Irritability (Psychiatric disorders) | 3 | 1
Memory Impairment (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT01847469/Prot_SAP_000.pdf